CLINICAL TRIAL: NCT02501486
Title: Inhalation or Nasal Corticosteroids and Prevalence of Hypothalamic-pituitary-adrenal Axis Suppression in HIV-infected Patients
Brief Title: Inhalation/Nasal Corticosteroids and Prevalence of Hypothalamic-pituitary-adrenal (HPA) Axis Suppression in Human Immunodeficiency Virus (HIV)-Patients
Acronym: Incorporate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: AIDS Fonds (Other); OLVG (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL51711.091.14
Record Dates: First submitted 2015-06-02; First posted 2015-07-17 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Adrenal Insufficiency
Keywords: adrenal insufficiency; adverse drug reaction; corticosteroid
MeSH Terms: conditions — Adrenal Insufficiency; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACTH stimulation test (Other): this is a single arm study. An ACTH-stimulation test will be done
  Interventions: Other: ACTH stimulation test

INTERVENTIONS:
Other: ACTH stimulation test — An ACTH stimulation test will be done

SUMMARY:
Rationale: Case reports describe suppression of the hypothalamic-pituitary-adrenal (HPA) axis caused by local corticosteroids, most often with inhalation corticosteroids. The exact prevalence is not known. Early recognition is important, because suppression of the HPA-axis can lead to significant morbidity and mortality. Suppression of the HPA axis might occur more often when a Cytochrome P450 3A4 (CYP3A4) inhibitor, e.g. ritonavir, is used next to the local corticosteroid, a combination often used by human immunodeficiency virus (HIV)-patients. Cortisol can be determined in hair. This non-invasive analysis could help in diagnosis of suppressed HPA-axis.

Research questions:

Primary objective:

1. How often do inhalation or nasal corticosteroids lead to suppression of the HPA- axis in HIV-treated patients?

   Secondary objectives:
2. Are other variables associated with the HPA-axis suppression?
3. Are cortisol measurements in hair as reliable as serum cortisol or an Adrenocorticotropic hormone (ACTH) stimulation test to diagnose suppression of the HPA axis? Study design: cross-sectional explorative study Study population: adults treated for HIV and using an inhalation or nasal corticosteroid.

Intervention: an ACTH stimulation test, cortisol measurements in blood and hair.

Main study parameters/endpoints:

Proportions of persons with a low morning plasma cortisol or low cortisol after an ACTH stimulation test. Correlation between cortisol in plasma and hair cortisol.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Each person will be screened with a history and a short physical examination. A venous cannula will be inserted for obtaining blood for the plasma cortisol and for the ACTH stimulation test. An ACTH stimulation test has no major complications. A piece of hair is cut for cortisol hair analysis. The risks and burden are minimal, while the future benefits could be great since suppression of the endogenous HPA- axis can be associated with morbidities like hypertension or osteoporosis and can even lead to an adrenal crisis when the local corticosteroid is stopped.

ELIGIBILITY:
Inclusion Criteria:

* Receive a treatment for HIV-infection
* > 18 years old
* Current usage of inhalation or nasal corticosteroids, for at least two weeks
* Willing to give informed consent

Exclusion Criteria:

* adrenal insufficiency
* Concurrent use of topical corticosteroids, usage of oral corticosteroids in the last three months. Intramuscular or intra-articular corticosteroid injections in the last year.
* Contra-indications for tetracosactide: allergy for tetracosactide, Cushings's syndrome, refractory heart failure, peptic ulcer, acute psychosis, adrenogenital syndrome
* If the patient ever had an ACTH-stimulation test before
* Pregnant female or breast-feeding female.
* Use of oral contraceptives, since these can heighten the cortisol-binding globulin
* Exclusion criterion for the cortisol measurements in hair: baldness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-01 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
the percentage of participants with a morning serum cortisol below 80 nmol/L in morning or below 550 nmol/L after Adrenocorticotropic (ACTH) stimulation test | baseline
  these are the persons with hypothalamic-pituitary-adrenal (HPA) -axis suppression

SECONDARY OUTCOMES:
Difference in percentage of HPA-axis suppression in participants who use a Cytochrome P450 3A4 (CYP3a4) inhibitor (ritonavir or cobicistat) versus percentage of HPA-axis suppression in participants who don't use a booster | baseline
  HPA-axis suppression is described in outcome 1. If the investigators have enough data the following will also be analysed: duration of usage of inhalation/nasal corticosteroids and use of systemical corticosteroid before (never versus ever used).
Percentage of HPA-axis suppression stratified by type of corticosteroid | baseline
  HPA-axis suppression is described in outcome 1. If the investigators have enough data the following will also be analysed: duration of usage of inhalation/nasal corticosteroids and use of systemical corticosteroid before (never versus ever used).
Difference in percentage of HPA-axis suppression in persons who use a high dose of corticosteroids versus a low dose of corticosteroids | baseline
Cortisol measurements in hair to diagnose HPA-axis suppression, in comparison with serum cortisol or an ACTH stimulation test | baseline
  hair cortisol measurements are given in pg/mg hair.

CONTACTS AND LOCATIONS:
Overall Officials: David Burger, Prof, Principal Investigator — Radboud UMC Pharmacy
Locations (2):
- Netherlands (2):
  - Onze lieve vrouw Gasthuis, Amsterdam
  - Radboud UMC, Nijmegen

REFERENCES:
- [Derived] Besemer F, Kramers C, Brinkman K, Hermus ARMM, van Herwaarden AE, Burger DM. Hypothalamic-pituitary-adrenal axis suppression by inhaled or nasal corticosteroids in HIV-infected patients. Int J Clin Pharm. 2020 Apr;42(2):347-350. doi: 10.1007/s11096-020-00995-5. Epub 2020 Mar 5. PMID 32140912